CLINICAL TRIAL: NCT07053137
Title: Comparing Efficacy and Safety of Telitacicept and Belimumab in Systemic Lupus Erythematosus: A Retrospective Multicenter Cohort Study
Brief Title: A Comparative Study of the Efficacy and Safety of Telitacicept and Belimumab in the Treatment of Systemic Lupus Erythematosus Involving Multiple Units, Based on Previous Data.
Status: Active, not recruiting | Type: Observational
Sponsor: Yipeng Liu (Other)
Collaborators: Renmin Hospital of Wuhan University (Other); Affiliated Hospital of Shandong University of Traditional Chinese Medicine (Other); Beijing Friendship Hospital (Other)
Responsible Party: Sponsor-Investigator, Yipeng Liu, Clinical Professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2025(101)
Record Dates: First submitted 2025-06-13; First posted 2025-07-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-07

CONDITIONS: Systemic Lupus Erythematosus; Telitacicept; Belimumab; Efficacy and Safety
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The Belimumab group: The participants in the study had previously used belimumab as a therapeutic drug.
- The Telitacicept group: The participants in the study had previously used telitacicept as a therapeutic drug.

SUMMARY:
The objective of this observational study is to compare the efficacy and safety of tixocutibine and belizumab in the treatment of systemic lupus erythematosus in patients aged 18-65 years with systemic lupus erythematosus. The main question it aims to answer is: In the overall population of systemic lupus erythematosus: What is the response rate (SRI-4) of the two drugs in treating systemic lupus erythematosus? Which drug has better efficacy and safety? This study is a retrospective study. The participants will not receive any treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18 - 65 years old;
* Meets the revised SLE classification criteria of the American College of Rheumatology in 1997 or the SLE diagnostic classification criteria issued by EULAR/ACR in 2019;
* SELENA-SLEDAI score of at least 8 points (clinical symptoms of no less than 6 points, excluding positive anti-double-stranded DNA (anti-dsDNA) and low complement);
* Patients who have been using tofacitinib or belimumab for at least 12 weeks.

Exclusion Criteria:

* Having active central nervous system diseases;
* eGFR < 30 mL/min/1.73m², or undergoing hemodialysis or kidney transplantation;
* Pregnant women, or women planning to get pregnant in the near future while taking the medication, or lactating women;
* Participants who are simultaneously participating in other clinical studies;
* Patients who have received treatment with tixagrel or belimumab for less than 12 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The inclusion period is from March 1, 2021 to March 1, 2024. Patients who visited the First Affiliated Hospital of Shandong University Medical University, the Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Wuhan University People's Hospital, and the Department of Nephrology of Capital Medical University Affiliated Beijing Friendship Hospital for clinical diagnosis of systemic lupus erythematosus were included.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-11-30 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with a Systemic Lupus Erythematosus Response Index-4 (SRI-4) response | From baseline to the end of 1-year treatment period
  1. The SELENA-SLEDAI score decreased by ≥ 4 points compared to the baseline;
  2. And there were no new BILAG-assessed grade A organs or ≤ 2 new BILAG-assessed grade B organs compared to the baseline;
  3. And the overall physician assessment (PGA) did not deteriorate (an increase of < 0.30 points compared to the baseline).

SECONDARY OUTCOMES:
Proportion of Participants with Stable SLEDAI and PGA Scores | From baseline to the end of 1-year treatment period
  The percentage of study participants whose SLEDAI score decreased by at least 4 points and whose PGA did not worsen.
The proportion of participants in the study who had their hormone dosage reduced | From baseline to the end of 1-year treatment period
  The ratio of study participants whose prednisone dose was reduced by ≥25% or ≤7.5 mg/day compared to the baseline at 44-48 weeks.
The time of recurrence occurrence | From baseline to the end of 1-year treatment period
  The time of the first recurrence or the first severe recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No